CLINICAL TRIAL: NCT04129047
Title: Shade Matching of Omnichroma (One Shade Universal Composite) Versus a Microhybrid Composite in Class V Restorations. A Randomized Clinical Trial
Brief Title: Shade Matching of Omnichroma (One Shade Universal Composite) Versus a Microhybrid Composite in Class V Restorations.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Mohamed Aly Aref, Resident, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OPER 3-7-1
Record Dates: First submitted 2019-10-12; First posted 2019-10-16 (Actual); Last update posted 2019-10-16 (Actual); Status verified 2019-10

CONDITIONS: Class V Restorations

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Omnichroma (one shade universal) composite by Tokuyama (Experimental): class V cavities will be made under isolation. Omnichroma (one shade universal) composite by Tokuyama will be placed according to guidelines.
  Interventions: Drug: Omnichroma (one shade universal) composite by Tokuyama
- A microhybrid composite Z250 (3 M ESPE, St. Paul, MN, USA) (Active Comparator): class V cavities will be made under isolation. A microhybrid composite Z250 (3 M ESPE, St. Paul, MN, USA) will be placed according to guidelines.
  Interventions: Drug: A microhybrid composite Z250 (3 M ESPE, St. Paul, MN, USA

INTERVENTIONS:
Drug: Omnichroma (one shade universal) composite by Tokuyama — Omnichroma is a single shade composite that is intended to have a color blending potential. It eliminates the shade matching procedures and makes it easier to avoid individual errors in shade matching in composite restorations.
  Arms: Omnichroma (one shade universal) composite by Tokuyama
Drug: A microhybrid composite Z250 (3 M ESPE, St. Paul, MN, USA — a multiple shade universal composite that needs prior shade selection procedure
  Arms: A microhybrid composite Z250 (3 M ESPE, St. Paul, MN, USA)

SUMMARY:
Background Resin composites are effective in restoring damaged teeth due to their good esthetics, high surface gloss, and clinically acceptable wear resistance1. One of the most challenging tasks a dentist has to confront in daily practice is matching the color of composite restorations used in anterior teeth2.

Problem The shade selection is carried out subjectively with a visual shade guide and generally under inadequate light conditions, which can lead to errors in color perception3. The presence of discrepancies between the classic shade guides and the actual shade of composite makes that task more difficult.4. Not only that, but there was also mismatch between composite shades and the proprietary shade guides included with the composite kits 5. A mock-up should be performed as a trial to assist in shade selection and ensure the predictability of the esthetic result in restorative treatment6.

Rationale Shade matching has been a time consuming procedure. Recommendations were made to make customized shade guides of the used composite material for more predictable results7. Manufacturers have been aiming at providing materials with a blending effect; taking on the color appearance from surrounding tooth structure 8. Introduction of Omnichroma by Tokuyama is aiming at eliminating the shade taking procedure by providing a single shade universal composite that is designed to blend with the surrounding tooth structure without the need for a shade matching procedure.

Aim The aim of this study is to evaluate the shade matching ability of a new single shade composite (Omnichroma; Tokuyama) compared to a conventional multiple shade microhybrid composite in the restoration of class V restorations using USPHS criteria

DETAILED DESCRIPTION:
Background and rationale:

Research question:

In class V restorations will there be a difference in shade matching between Omnichroma (one shade) universal composite and a microhybrid (multiple shade) universal composite?

Statement of the problem:

The shade selection is carried out subjectively with a visual shade guide and generally under inadequate light conditions, which can lead to errors in color perception. The presence of discrepancies between the classic shade guides and the actual shade of composite makes that task more difficult. Not only that, but there was also mismatch between composite shades and the proprietary shade guides included with the composite kits. A mock-up should be performed as a trial to assist in shade selection and ensure the predictability of the esthetic result in restorative treatment.

Rationale for conducting the research:

Shade matching has been a time-consuming procedure. Recommendations were made to make customized shade guides of the used composite material for more predictable results. Manufacturers have been aiming at providing materials with a blending effect; taking on the color appearance from surrounding tooth structure. Introduction of Omnichroma by (Tokuyama Dental, Tokyo, Japan) is aiming at eliminating the shade taking procedure by providing a single shade universal composite that is designed to blend with the surrounding tooth structure without the need for a shade matching procedure.

Review of literature:

In 2004, Nahri compared the clinical efficacy of Z250 (3M, Saint Paul, MN, USA) with Z100 (3M, Saint Paul, MN, USA) in class III and class V restorations. A total of 148 restorations were placed by different dentists. The study used modified USPHS criteria to evaluate the restorations at baseline and for one year. Color match, along with marginal adaptation, discoloration, and anatomic form were evaluated using specified criteria. Baseline evaluation was done after one week from restoration placement. At baseline, 70% of the Z250 restorations were rated as Alpha regarding color-match compared to 62% of the Z100 restorations. It was concluded that there was no significant difference between the two materials and that both can be used in class V restorations.

A study by Sakrana compared between the clinical performance of Palfique Estelite,( Tokuyama Corp., Tokyo, Japan) resin composite and Palfique Toughwell (Tokuyama Corp., Tokyo, Japan) Resin Composite in anterior class V restorations. Both are minifilled composites with Palfique Estelite indicated for anterior restorations and Palfique Toughwell indicated for both anterior and posterior ones. Seventy eight class V cavities were restored using Palfique Estellite and eighty two were restored with Palfique Toughwell. Both groups were examined immediately after polishing (baseline), after 6 months, and after 1 year. Both showed 100% color match of rating Alpha (USPHS criteria) at baseline. At 6 months, 100 % of Palfique Estelite restorations were still rated as Alpha, while only 90% of the Palfique Toughwell restorations were still rated as Alpha. It was shown that Palfique Toughwell had more color change after one year. Only 70% were rated as Alpha regarding color match after one year. However, the difference was not significant and both materials prove to be reliable in class V restorations.

Another study by Paravina found color differences between same shades of 2 microhybrid composite when placed in specimens of different surrounding color or different size. They used specimens of 2 composite shades placed circumferentially. The outer ring was using the darker composite and the inner was the lighter. Palfique Estellite (Tokuyama, Tokyo, Japan) composite of shade C2 was used as the darker outer composite. Lighter shades (A2 and B2) of Palfique Estellite and Esthet-X (Dentsply/Caulk, Milford, DE) were used in the inner part. Multiple diameters (2,4,6) of the inner part were used. In addition to that, single composite specimens were prepared from the same shades for comparison. It was found that the same shades of composite appeared differently when placed in different diameters. Also, when there was less color difference between inner and outer disks, more color match is achieved. This led to a conclusion that composites can have a blending effect. This blending effect increased with decreased restoration size, decreased color difference, and translucency of the used composite.

Mourouzis compared the blending effect of three commercially available composites in vitro, microhybrid GC Gradia Direct Anterior (GC Corporation, Tokyo, Japan), microfilled Clearfil Majesty Esthetic (Kuraray Medical Inc., Tokyo, Japan), and nanofilled IPS Empress Direct (Ivoclar Vivadent, Shaan, Liechtenstein). The study was conducted on extracted teeth. Shade was taken for the teeth using a spectrophotometer. The teeth were sectioned vertically and restored using the three composite materials of the designated shade. The restorations were made using a prefabricated mold. The shade was taken afterwards and compared to that of intact teeth. Results were that all composite restorations had color differences with intact teeth. However, this difference was not visible by human eye and it was concluded that a color difference of ΔΕ<3.3 was considered clinically acceptable It was stated that the properties of the composite material have a drastic effect over esthetics. The Ivoclar group demonstrated the most color difference among the 3 groups.

McLaren et al introduced a technique using calibrated photography and photoshop for shade analysis. Digital photographs were taken in Raw format using polarizing filters and a gray card. The cross-polarizing filter is used for eliminating glare. The gray card is used to calibrate exposure in Adobe Camera Raw (which comes in adjunction with Adobe Photoshop to compensate for exposure differences between different camera-models. The authors provided recommended camera settings for standardization of images. L, A, and B values were calculated using digital color meter in photoshop and compared to those of shade tabs for shade selection. The authors claimed this technique to be effective, useful, and accurate in shade analysis.

In 2019, Paravina et al compared between color adjusting potential of 5 commercially available universal composites namely Omnichroma (Tokuyama Dental, Tokyo, Japan), Filtek Supreme Ultra (3M, Saint Paul, MN), TPH Spectra (Dentsply Caulk, Milford, DE), Herculite Ultra (Kerr Corporation, Orange, CA), and Tetric Evoceram (Ivoclar Vivadent, Amherst, NY) in vitro. Single and dual specimens were prepared. Single specimens were composed of the composite material alone and were compared to denture teeth. Dual specimens were composed of the restorative material placed in cavities prepared in acrylic teeth of different shades. Comparisons were made between denture teeth and single specimens and dual specimens. Comparisons were made visually and instrumentally. There was large color difference between single specimens and Denture teeth. However, dual specimens showed more color match. This was most pronounced in Omnichroma. It was concluded that Omnichroma had the most color adjusting potential. This means that it had a great color difference between single specimens and denture teeth. It also had the greatest color match in dual specimens.

6b. Explanation for choice of comparators:

Micro-hybrid composite was chosen as a comparator because it's considered a universal composite to be used in anterior and posterior restorations. It has high filler content along with good surface polish and color stability. Also according to a recent study, micro-hybrid composite showed excellent color match and color stability compared to nano-filled composite in five-years follow-up.

Interventions:

Patients attending at the Conservative and Esthetic Dentistry Department Clinic will be screened. Those who meet the study inclusion criteria will be recruited. They will be informed with the study and an informed consent will be signed if they approve.

First Periodontal treatment will be made and oral hygiene instructions will be enforced. Shade taking procedure will be done visually using customized composite shade tabs for more accuracy. Shade will be confirmed using cross-polarized photography and image analysis using a digital color meter (Adobe Photoshop).

Once the shade is confirmed, the operator will start rubber-dam isolation and cavity preparation using a round bur. Remaining caries will be excavated by a sharp excavator. A 1mm bevel will be prepared in enamel margins.

Selective enamel etching will be done and a universal adhesive will be applied to both enamel and dentin. After solvent evaporation, the bonding agent will be cured for 20 seconds. The operator will be blinded to the material to be used till the placement of the restoration to avoid bias. According to the concealed envelope, the tooth will be assigned to one of both treatment groups. Composite will be placed incrementally and light cured for 20 seconds using 3M Elipar DeepCure-S LED Curing Light (3M, Saint Paul, MN, USA)

Post curing will be done using Glycerin to decrease the oxygen inhibited layer. Finishing will be done using yellow and white finishing stones Intensiv (Intensiv SA, Montagnola, Switzerland). More finishing and polishing will be done using (Enhance and Pogo (Dentsply Sirona). Rubber-dam will be removed and patients will be recalled for baseline evaluation after one week to allow for rehydration.

The assessor will be blinded to both treatment groups. She will give the restorations a score using Modified USPHS score. Calibrated photographs will be taken using cross polarizing filters and a gray card for image analysis using Photoshop.

Recall appointments will be after 3 months and 6 months. Same evaluation will be made to assess color stability.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with carious class V lesions
2. Non-carious cervical abfraction lesions
3. Young adult Males or female
4. Good oral hygiene
5. Co-operative patients approving to participate in the study

Exclusion Criteria:

1. Patients with a compromised medical history.
2. Severe or active periodontal disease
3. Severe medical complications
4. Erosive lesions
5. Lack of compliance and rampant caries

Ages: 15 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 38 (Estimated)
Dates: Start 2019-07-20 (Actual); Primary Completion 2020-04 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Shade matching (visually and using image analysis) | Baseline after 1 week
  To evaluate the shade matching ability of the newly introduced single shade composite compared to a conventional multiple shade micro hybrid composite. Assessment will be done visually using Modified USPHS Criteria and by image analysis. Image analysis will be done by comparing LAB values using Adobe Photoshop

SECONDARY OUTCOMES:
Color stability (visually and using image analysis) | Color stability between baseline, 3 months and 6 months
  To evaluate the color stability of the newly introduced single shade composite compared to a conventional multiple shade micro hybrid composite. Assessment will be done visually using Modified USPHS Criteria and by image analysis. Image analysis will be done by comparing LAB values using Adobe Photoshop

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sakrana AA, Tanoue N, Kawasaki K, Matsumura H. One-year clinical evaluation of two composite materials used for anterior class V restorations. J Oral Rehabil. 2004 Oct;31(10):985-90. doi: 10.1111/j.1365-2842.2004.01333.x. PMID 15387839
- [Background] Bayne SC, Heymann HO, Swift EJ Jr. Update on dental composite restorations. J Am Dent Assoc. 1994 Jun;125(6):687-701. doi: 10.14219/jada.archive.1994.0113. PMID 8014334
- [Background] Ferracane JL. Resin composite--state of the art. Dent Mater. 2011 Jan;27(1):29-38. doi: 10.1016/j.dental.2010.10.020. Epub 2010 Nov 18. PMID 21093034
- [Background] Folwaczny M, Loher C, Mehl A, Kunzelmann KH, Hickel R. Class V lesions restored with four different tooth-colored materials--3-year results. Clin Oral Investig. 2001 Mar;5(1):31-9. doi: 10.1007/s007840000098. PMID 11355096
- [Background] Fondriest J. Shade matching in restorative dentistry: the science and strategies. Int J Periodontics Restorative Dent. 2003 Oct;23(5):467-79. PMID 14620121
- [Background] Hall NR, Kafalias MC. Composite colour matching: the development and evaluation of a restorative colour matching system. Aust Prosthodont J. 1991;5:47-52. PMID 1812939
- [Background] Kim HS, Um CM. Color differences between resin composites and shade guides. Quintessence Int. 1996 Aug;27(8):559-67. PMID 9161260
- [Background] Lee YK, Yu B, Lee SH, Cho MS, Lee CY, Lim HN. Shade compatibility of esthetic restorative materials--A review. Dent Mater. 2010 Dec;26(12):1119-26. doi: 10.1016/j.dental.2010.08.004. Epub 2010 Sep 15. PMID 20832851
- [Background] McLaren EA, Figueira J, Goldstein RE. A Technique Using Calibrated Photography and Photoshop for Accurate Shade Analysis and Communication. Compend Contin Educ Dent. 2017 Feb;38(2):106-113. PMID 28156124
- [Background] Mourouzis P, Koulaouzidou EA, Palaghias G, Helvatjoglu-Antoniades M. Color match of resin composites to intact tooth structure. J Appl Biomater Funct Mater. 2015 Oct 16;13(3):e259-65. doi: 10.5301/jabfm.5000228. PMID 26108430
- [Background] Narhi TO, Tanner J, Ostela I, Narva K, Nohrstrom T, Tirri T, Vallittu PK. Anterior Z250 resin composite restorations: one-year evaluation of clinical performance. Clin Oral Investig. 2003 Dec;7(4):241-3. doi: 10.1007/s00784-003-0231-6. Epub 2003 Sep 18. PMID 14505071
- [Background] Paravina RD, Westland S, Kimura M, Powers JM, Imai FH. Color interaction of dental materials: blending effect of layered composites. Dent Mater. 2006 Oct;22(10):903-8. doi: 10.1016/j.dental.2005.11.018. Epub 2005 Dec 27. PMID 16378637
- [Background] Paravina RD, Kimura M, Powers JM. Color compatibility of resin composites of identical shade designation. Quintessence Int. 2006 Oct;37(9):713-9. PMID 17017633
- [Background] Pereira Sanchez N, Powers JM, Paravina RD. Instrumental and visual evaluation of the color adjustment potential of resin composites. J Esthet Restor Dent. 2019 Sep;31(5):465-470. doi: 10.1111/jerd.12488. Epub 2019 May 16. PMID 31095870
- [Background] Ruschel VC, Martins MV, Bernardon JK, Maia HP. Color Match Between Composite Resin and Tooth Remnant in Class IV Restorations: A Case Series. Oper Dent. 2018 Sep/Oct;43(5):460-466. doi: 10.2341/17-132-S. Epub 2018 Mar 16. PMID 29547347
- [Background] Strnad, G. et al. (2015) 'Effect of Curing, Finishing and Polishing Techniques on Microhardness of Composite Restorative Materials', Procedia Technology, 19, pp. 233-238. doi: https://doi.org/10.1016/j.protcy.2015.02.034.
- [Background] Tuncer S, Demirci M, Oztas E, Tekce N, Uysal O. Microhybrid versus nanofill composite in combination with a three step etch and rinse adhesive in occlusal cavities: five year results. Restor Dent Endod. 2017 Nov;42(4):253-263. doi: 10.5395/rde.2017.42.4.253. Epub 2017 Aug 21. PMID 29142873